CLINICAL TRIAL: NCT00709371
Title: A Phase IIB, Multi-Center, Dose-Parallel, Randomized, Double-Blind, Monotherapy and Placebo-Controlled Safety and Efficacy Study of Zonisamide SR Plus Bupropion SR Combination Therapy in Subjects With Obesity
Brief Title: Zonisamide SR Plus Bupropion SR Combination Therapy in Subjects With Obesity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZB-202
Record Dates: First submitted 2008-06-29; First posted 2008-07-03 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: obesity; zonisamide; bupropion
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Combination tablet containing Zonisamide SR placebo plus bupropion SR placebo SR = Sustained Release
  Interventions: Drug: Zonisamide SR placebo/ bupropion SR placebo
- Bupropion 360 (Active Comparator): Combination tablet containing Zonisamide SR placebo plus bupropion SR 360 mg/day; SR = Sustained Release
  Interventions: Drug: Zonisamide SR placebo/ bupropion SR 360 mg/day
- Zonisamide 120 (Active Comparator): Combination tablet containing Zonisamide SR 120 mg/day plus bupropion SR placebo; SR = Sustained Release
  Interventions: Drug: Zonisamide SR 120 mg/day/ bupropion SR placebo
- Zonisamide 360 (Active Comparator): Combination tablet containing Zonisamide SR 360 mg/day plus bupropion SR placebo; SR = Sustained Release
  Interventions: Drug: Zonisamide SR 360 mg/day/ bupropion SR placebo
- Zonisamide 120/Bupropion 360 (Experimental): Combination tablet containing Zonisamide SR 120 mg/day plus bupropion SR 360 mg/day; SR = Sustained Release
  Interventions: Drug: Zonisamide SR 120 mg/day/ bupropion SR 360 mg/day
- Zonisamide 360/Bupropion 360 (Experimental): Combination tablet containing Zonisamide SR 360 mg/day plus bupropion SR 360 mg/day; SR = Sustained Release
  Interventions: Drug: Zonisamide SR 360 mg/day/ bupropion SR 360 mg/day

INTERVENTIONS:
Drug: Zonisamide SR placebo/ bupropion SR placebo — 2 placebo combination tablets twice daily for 16 weeks (maintenance period)
  Arms: Placebo
Drug: Zonisamide SR placebo/ bupropion SR 360 mg/day — 2 placebo and bupropion SR 90 mg combination tablets, twice daily for 16 weeks (maintenance period)
  Arms: Bupropion 360
Drug: Zonisamide SR 120 mg/day/ bupropion SR placebo — 2 zonisamide SR 30 mg and placebo combination tablets, twice daily for 16 weeks (maintenance period)
  Arms: Zonisamide 120
Drug: Zonisamide SR 360 mg/day/ bupropion SR placebo — 2 zonisamide SR 90 mg and placebo combination tablets, twice daily for 16 weeks (maintenance period)
  Arms: Zonisamide 360
Drug: Zonisamide SR 120 mg/day/ bupropion SR 360 mg/day — 2 zonisamide SR 30 mg and bupropion SR 90 mg combination tablets, twice daily for 16 weeks (maintenance period)
  Arms: Zonisamide 120/Bupropion 360
Drug: Zonisamide SR 360 mg/day/ bupropion SR 360 mg/day — 2 zonisamide SR 90 mg and bupropion SR 90 mg combination tablets, twice daily for 16 weeks (maintenance period)
  Arms: Zonisamide 360/Bupropion 360

SUMMARY:
The purpose of this study is determine if the combination of zonisamide SR and bupropion SR are is more effective than either drug given alone or placebo in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects, 18 to 65 years of age
* Have body mass index (BMI) ≥ 30 kg/m2 and ≤ 45 kg/m2 for subjects with uncomplicated obesity, and BMI of ≥ 27 kg/m2 and ≤ 45 kg/m2 for subjects with obesity and dyslipidemia and/or controlled hypertension
* Non-smoker and no use of tobacco or nicotine products for at least 6 months prior to screening
* Normotensive (systolic ≤140 mm Hg; diastolic ≤90 mm Hg). Anti-hypertensive medications are allowed with the exception of adrenergic blockers and clonidine. Medical regimen must be stable for at least 6 weeks prior to randomization
* Triglycerides <400 mg/dL. Medications for treatment of dyslipidemia are allowed with the exception of cholestyramine and cholestypol as long as medical regimen has been stable for at least 6 weeks prior to randomization
* No clinically significant laboratory abnormalities
* Negative urine drug screen
* Negative serum pregnancy test in women of child-bearing potential
* Women of child-bearing potential must be non-lactating, and agree to use acceptable contraception throughout the study period and for 30 days after discontinuation of study drug
* Able to comply with all required study procedures and schedule
* Able to speak and read English
* Willing and able to give written informed consent

Exclusion Criteria:

* Obesity of known endocrine or genetic origin (e.g., untreated hypothyroidism, Cushing's syndrome, polycystic ovary syndrome)
* Serious medical condition
* History of malignancy within the previous 5 years, with exception of non-melanoma skin cancer or surgically cured cervical cancer.
* History of suicide attempt or serious psychiatric illness
* History of Major Depressive Disorder within the past 2 years
* In need of medications for the treatment of a psychiatric disorder (with the exception of short-term insomnia) within the previous 6 months prior to randomization
* Type I or Type II diabetes
* History of alcohol or drug abuse or dependence as determined by the Investigator within 1 year prior to randomization
* History of surgical or device (e.g. gastric banding) intervention for obesity
* History of seizures or predisposition to seizures
* History of hypersensitivity to sulfonamides ("sulfa"), bupropion, or zonisamide
* History of treatment with bupropion SR (Wellbutrin, Zyban) or zonisamide (Zonegran) within previous 12 months
* History of nephrolithiasis (renal calculi)
* Loss or gain of more than 4.0 kg within 3 months prior to randomization
* Women of child bearing potential not adhering to a medically acceptable form of contraception
* Pregnant or breast-feeding women or planning to become pregnant during the study period or within 30 days of discontinuing study drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 729 (Actual)
Dates: Start 2008-07; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percentage change in total body weight | from baseline to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Acampora, MD, Principal Investigator — Internal Medicine Associates of Charlotte; Caroline Apovian, MD, Principal Investigator — Nutrition and Weight Management Center; James Bergthold, MD, Principal Investigator — Summit Research Network (Oregon), Inc.; Joseph Cleaver, MD, Principal Investigator — The Cooper Institute; Adnan Dahdul, MD, Principal Investigator — FutureCare Studies; Ken Fujioka, MD, Principal Investigator — Nutrition and Metabolic Research; Jeffrey Geohas, MD, Principal Investigator — Radiant Research, Chicago; Mark Graves, MD, Principal Investigator — Welborn Clinic; Alok Gupta, MD, Principal Investigator — Pennington Biomedical Research Center; Wayne Harper, MD, Principal Investigator — Wake Research Associates, LLC; Jonathan Henry, MD, Principal Investigator — Summit Research Network (Michigan), Inc.; Diane Krieger, MD, Principal Investigator — Miami Research Associates; Michael Levy, MD, Principal Investigator — Behavioral Medical Research; Raymond Plodkowski, MD, Principal Investigator — Center for Nutrition and Metabolic Disorders, University of Nevada School of Medicine; Domenica Rubino, MD, Principal Investigator — Washington Center for Weight Management and Research; Stan Self, MD, Principal Investigator — SelfCenter, PC; Diane Smith, MD, Principal Investigator — CSRA Partners in Health, Inc.; Timothy Smith, MD, Principal Investigator — Mercy Research; Claire Waltman, MD, Principal Investigator — Summit Research Network (Seattle), LLC; Holly Wyatt, MD, Principal Investigator — Center for Human Nutrition/UCD
Locations (20):
- United States (20):
  - SelfCenter, PC, Fairhope, Alabama
  - Nutrition and Metabolic Research, La Jolla, California
  - Center for Human Nutrition/UCD, Denver, Colorado
  - Miami Research Associates, Miami, Florida
  - CSRA Partners in Health, Inc., Augusta, Georgia
  - Radiant Research, Chicago, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Nutrition and Weight Management Center, Boston Medical Center, Boston, Massachusetts
  - FutureCare Studies, Springfield, Massachusetts
  - Summit Research Network (Michigan), Inc., Farmington Hills, Michigan
  - Mercy Health Research, St Louis, Missouri
  - Center for Nutrition and Metabolic Disorders, University of Nevada School of Medicine, Reno, Nevada
  - Behavioral Medical Research, Staten Island, New York
  - Internal Medicine Associates of Charlotte, Charlotte, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Summit Research Network (Oregon), Inc., Portland, Oregon
  - The Cooper Institute, Dallas, Texas
  - Washington Center for Weight Management and Research, Arlington, Virginia
  - Summit Research Network (Seattle), LLC., Seattle, Washington